CLINICAL TRIAL: NCT01142674
Title: Prospective Collection of Data in Pts With Peripheral T-Cell Lymphoma: PTCL,NOS;AITL; Extranodal NK/T-cell;Enteropathy-type; Hepatosplenic γ-δ; Subcutaneous Panniculitis-like; ALCL,Primary Systemic Type. By the Intl. T-Cell Lymphoma Project
Brief Title: T-Cell Project: Prospective Collection of Data in Patients With Peripheral T-Cell Lymphoma
Status: Completed | Type: Observational
Sponsor: Associazione Angela Serra per la ricerca sul cancro (Other)
Collaborators: Fondazione Italiana Linfomi - ETS (Other); INTERNATIONAL T-CELL NON-HODGKIN'S LYMPHOMA STUDY GROUP (Unknown)
Responsible Party: Sponsor
Other Study IDs: T-Cell Project
Record Dates: First submitted 2010-06-10; First posted 2010-06-11 (Estimated); Last update posted 2019-07-08 (Actual); Status verified 2019-07

CONDITIONS: Lymphoma, T-Cell, Peripheral
Keywords: Lymphoma, T-Cell, Peripheral; Prognosis; Outcome; International Cooperation; Biological Characteristics; Heterogeneity; Rare Diseases
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral; Rare Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Formalin-fixed tissue for central diagnostic pathology review
Oversight: Data Monitoring Committee: No

SUMMARY:
The designed study follows up the retrospective previous one by the International T-cell Non-Hodgkin's Lymphoma Study Group (International Peripheral T-Cell Lymphoma Project).

It is designed as a prospective collection of information potentially useful to predict the prognosis of newly diagnosed patients with the more frequent subtypes of Peripheral T-cell lymphoma (Peripheral T-cell lymphoma unspecified and Angioimmunoblastic T-cell lymphoma) and to better define clinical characteristics and outcome of the more uncommon subtypes

DETAILED DESCRIPTION:
Peripheral T-cell lymphomas (PTCLs) comprise a heterogeneous group of neoplasms that are derived from post-thymic lymphoid cells at different stages of differentiation with different morphological patterns, phenotypes, and clinical presentations. PTCLs are highly diverse, reflecting the diverse cells from which they can originate. Peripheral T-Cell Lymphomas account for 5-10% of all lymphoproliferative disorders in the Western hemisphere, with an overall incidence of 0.5-2 per 100,000 per year, and have a striking epidemiological distribution, with higher incidence in Asia.

The clinical features of PTCLs are extremely heterogeneous. PTCLs express even more clinical diversity than B-cell NHLs, and there is a close, though not absolute, relationship between some unusual clinical features and certain histological subtypes. Despite efforts to transferring to patients with T-cell lymphomas the most recent advances in the treatment of other subtypes of B-cell lymphomas, the prognosis of patients with PTCL is still poor an, unfortunately, the optimal therapy for PTCL is still unknown. The complete response rate is rather low, ranging from 40% to 50% with a median Relapse Free Survival (RFS) of 2-3 years. As a consequence of the aggressiveness of the disease and of the low efficacy of available salvage treatments, Overall Survival (OS) is also short and the long-term survival rate is lower than 10% in many series.

To better define the clinical outcome of PTCL-NOS, the Intergruppo Italiano Linfomi (IIL, now Fondazione Italiana Linfomi, FIL) performed a large study on 385 patients diagnosed and treated in the 1990s and defined a prognostic model specifically devised for patients with this uncommon disease (Gallamini, A. et al Blood, 2004. 103(7): p. 2474-9). In addition to defining a prognostic model specifically devised for PTCL-NOS, the FIL study confirms the relevance of research on series of clearly defined cases in order to the development of rationally designed and potentially more-efficacious treatment modalities. More recently, the role of biological features of the disease is emerging as an important issue not only for understanding its pathogenesis but also for prognosis and for addressing specific biologic targets altered in the neoplasia. Significant progress in the prognosis of PTCL can be expected from the novel, sophisticated, and powerful technologies of genomics and proteomics, which will allow more reliable subtyping of PTCL into distinct clinical groups characterized by different patterns of survival, as already demonstrated for some B-NHLs.

One common limitation of existing studies on prognosis of PTCL is their retrospective nature. Currently available data are based on analysis performed on series collected over a long period of time. This aspect is very important as it may introduce relevant biases in the collected series. First classification systems have changed dramatically over time and cases may have been defined in differently based on diagnosis year. Second some clinical or laboratory data which now are considered as prognostic relevant may have not been determined in older series of patients. Third in a retrospective analysis there is no guarantee that collected series are based on real consecutive cases. These are the reasons why we thought it would be useful to start a new study based on the prospective registration in a short period of time of patients with diagnosis of Peripheral T-cell lymphoma for whom it would be possible collect an exhaustive set of clinical data and biological information.

ELIGIBILITY:
Inclusion Criteria:

1. Previously-untreated patients with de novo diagnosis of peripheral T-cell or NK/T-cell lymphoma:

   * Peripheral T-cell lymphoma unspecified;
   * Peripheral T-cell lymphoma, lymphoepithelioid variant;
   * Peripheral T-cell lymphoma, T-zone variant ;
   * Peripheral T-cell lymphoma, parafollicular variant ;
   * Angioimmunoblastic T-cell lymphoma;
   * Nasal NK/T-cell lymphoma;
   * NK/T-cell lymphoma, nasal time;
   * Anaplastic large-cell lymphoma, T/null cell, ALK+, primary systemic type
   * Anaplastic large-cell lymphoma, T/null cell, ALK-, primary systemic type
   * Anaplastic large cell lymphoma, small cell variant, ALK+
   * Anaplastic large cell lymphoma, lymphohistiocytic variant, ALK+
   * Enteropathy- type T-cell lymphoma;
   * Hepatosplenic T-cell lymphoma;
   * Peripheral gamma-delta T-cell lymphoma;
   * Subcutaneous panniculitis-like T-cell lymphoma;
   * Unclassifiable peripheral T-cell Lymphoma
   * Unclassifiable NK-cell lymphoma
2. Age over 18
3. Tissue biopsies adequate for diagnosis and classification and available for centralized review
4. Clinical data including baseline information on disease localization and laboratory parameters at staging, features of treatment adopted and assurance of follow-up updating for at least 5 years are requested
5. Written informed consent

Exclusion Criteria:

1. Age < 18
2. Diagnosis of T-cell or NK-cell leukemia or proliferation and other than mature types including:

   * Adult T-cell leukemia/lymphoma;
   * Blastic NK-cell leukemia/lymphoma;
   * Aggressive NK-cell leukemia
   * T-cell large granular lymphocytic leukemia
   * T-cell large granular lymphocytic proliferation
   * NK-cell large granular lymphocytic proliferation
   * T-cell prolymphocytic leukemia
   * Precursor T-cell lymphoblastic leukemia/lymphoma
   * Mycosis fungoides;
   * Sézary syndrome;
   * Primary cutaneous ALCL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Previously-untreated patients with de novo diagnosis of peripheral T-cell or NK/T-cell lymphoma
Sampling Method: Non-Probability Sample
Enrollment: 1650 (Estimated)
Dates: Start 2006-09 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Overall Survival (OS) | 5 years

SECONDARY OUTCOMES:
Event Free Survival (EFS) | 5 years
Remission rate with initial therapy | End of front-line therapy
Progression Free Survival (PFS) | 5-years

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Federico, MD, Study Chair — Dip. Medicina Diagnostica - Università di Modena e Reggio Emilia, , Modena, IT; Julie M. Vose, MD, Study Chair — Nebraska Medical Center, Omaha, NE, USA; Emanuele Zucca, MD, Study Chair — IOSI/Oncology Institute of Southern Switzerland, Ospedale S. Giovanni - Bellinzona, CH; Joseph M Connors, MD, Study Chair — British Columbia Cancer Agency, Vancouver, CA; Steven M. Horwitz, MD, Study Chair — Memorial Sloan Kettering Cancer Center; Francine M. Foss, MD, Study Chair — Yale Cancer Center, New Haven, CT, USA; Pier Luigi Zinzani, MD, Study Chair — Istituto di Ematologia e Oncologia Medica "L. e A. Seragnoli", Policlinico Sant'Orsola, Bologna, IT; Silvia Montoto, MD, Study Chair — St. Bartholomew Hospital, London, UK; Aaron Polliack, MD, Study Chair — Sourasky Medical Center, Tel Aviv, IL; Stefano A. Pileri, MD, Study Chair — Università di Bologna, IT & Istituto Europeo di Oncologia, Milano, IT; Young H. Ko, MD, Study Chair — Samsung Medical Center, Seoul, KR
Locations (76):
- United States (8):
  - Stanford University Medical Center, Palo Alto, California
  - Yale Cancer Center, New Haven, Connecticut
  - St Louis Washington University, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - MD Anderson Cancer Center, Houston, Texas
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
- Argentina (3):
  - Hospital Italiano, La Plata, Buenos Aires
  - Hospital San Martìn, La Plata, Buenos Aires
  - Fundacion Fundaleu, Buenos Aires
- Brazil (2):
  - University of Campinas, Campinas, São Paulo
  - Santa Casa Medical School, São Paulo
- Hospital del Salvador SSMO, Santiago, Chile
- China (3):
  - Princess Margaret Hospital, Hong Kong
  - Queen Mary Hospital, Hong Kong
  - Tuen Mun Hospital, Hong Kong
- Hopital St Louis, Paris, France
- Israel (2):
  - Sheba Medical Center, Tel Aviv
  - Sourasky Medical Center, Tel Aviv
- Italy (41):
  - Presidio Spedali Civili, Brescia, BS
  - Azienda Ospedaliera S. Croce e Carle, Cuneo, CN
  - Presidio Ospedaliero Garibaldi-Nesima, Catania, CT
  - Azienda O.U. Vittorio Emanuele-Ferrarotto-S. Bambino, Catania, CT
  - Azienda Ospedaliera Pugliese-Ciaccio, Catanzaro, CZ
  - Ospedale Casa Sollievo della Sofferenza IRCCS, San Giovanni Rotondo, FG
  - Azienda Ospedaliera Vito Fazzi, Lecce, LE
  - Ospedale Civile, Civitanova Marche, Macerata
  - Azienda Ospedaliera Ospedali Riuniti Papardo-Piemonte, Messina, ME
  - Istituto Clinico Humanitas, Milan, MI
  - Istituto Scientifico Universitario San Raffaele, Milan, MI
  - Istituto Europeo di Oncologia, Milan, MI
  - Azienda Ospedaliera Ospedale Niguarda Ca' Franda, Milan, MI
  - Ospedale Madonna delle Grazie, Matera, Mount
  - Centro Oncologico Modenese, Modena, MO
  - Casa di Cura La Maddalena, Palermo, Pa
  - Istituto Oncologico Veneto, Padua, PD
  - Centro di Riferimento Oncologico, Aviano, Pordenone
  - Azienda Ospedaliera Bianchi-Melacrino-Morelli, Reggio Calabria, RC
  - Arcispedale S. Maria Nuova, Reggio Emilia, RE
  - Presidio Ospedaliero Umberto I, Nocera Inferiore, SA
  - Azienda Ospedaliera S. Giovanni Battista, Torino, TO
  - Istituto di Ematologia A & Seragnoli, Bologna
  - Ospedale Centrale di Bolzano, Bolzano
  - Ospedale A. Perrino, Brindisi
  - Ospedale Oncologico A. Businco, Cagliari
  - Azienda Ospedaliera Pugliese-Ciaccio, Catanzaro
  - Azienda Ospedaliera Universitaria Careggi, Florence
  - Ospedale Felettino, La Spezia
  - Fondazione Policlinico MaRe IRCCS, Milan
  - Azienda Ospedaliera Universitaria Federico II, Napoli
  - Azienda Ospedaliera Maggiore della Carità, Novara
  - Azienda Ospedaliero-Universitaria, Parma
  - Ospedale Santo Spirito, Pescara
  - Ospedale Guglielmo da Saliceto, Piacenza
  - Azienda Ospedaliera Universitaria Pisana, Pisa
  - Università La Sapienza, Roma
  - Ospedale S. Vincenzo, Taormina
  - Ospedale Moscati, Taranto
  - Azienda Ospedaliera S. Maria, Terni
  - Ospedale Civile SS. Giovanni e Paolo, Venezia
- Nacional Cancer Institute, Bratislava, Slovakia
- Samsung Medical Center, Seoul, South Korea
- Spain (2):
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitario, Salamanca
- Switzerland (3):
  - Kantonsspital, Aarau, Canton of Aargau
  - Ospedale S. Giovanni, Bellinzona, Canton Ticino
  - Kantonsspital St. Gallen, Sankt Gallen
- United Kingdom (7):
  - University Hospital Birmingham NHS Foundation Trust, Birmingham
  - Barths and The London NHS Trust, London
  - Guy's and St. Thomas NHS Foundation Trust, London
  - Christie Hospital NHS Foundation Trust, Manchester
  - Newcastle University, Newcastle upon Tyne
  - University of Southampton School of Medicine, Southampton
  - New Cross Hospital, Wolverhampton
- Hospital Maciel, Montevideo, Uruguay

IPD SHARING:
Plan to Share IPD: Yes
Preliminary analysis results will be made available during the study on the single population and separately for each subtype. Final results will be made available 6-12 months after the end of the study

REFERENCES:
- [Background] Harris NL, Jaffe ES, Diebold J, Flandrin G, Muller-Hermelink HK, Vardiman J, Lister TA, Bloomfield CD. World Health Organization classification of neoplastic diseases of the hematopoietic and lymphoid tissues: report of the Clinical Advisory Committee meeting-Airlie House, Virginia, November 1997. J Clin Oncol. 1999 Dec;17(12):3835-49. doi: 10.1200/JCO.1999.17.12.3835. PMID 10577857
- [Background] Jones D, O'Hara C, Kraus MD, Perez-Atayde AR, Shahsafaei A, Wu L, Dorfman DM. Expression pattern of T-cell-associated chemokine receptors and their chemokines correlates with specific subtypes of T-cell non-Hodgkin lymphoma. Blood. 2000 Jul 15;96(2):685-90. PMID 10887135
- [Background] Picker LJ, Weiss LM, Medeiros LJ, Wood GS, Warnke RA. Immunophenotypic criteria for the diagnosis of non-Hodgkin's lymphoma. Am J Pathol. 1987 Jul;128(1):181-201. PMID 3111266
- [Background] Cooke CB, Krenacs L, Stetler-Stevenson M, Greiner TC, Raffeld M, Kingma DW, Abruzzo L, Frantz C, Kaviani M, Jaffe ES. Hepatosplenic T-cell lymphoma: a distinct clinicopathologic entity of cytotoxic gamma delta T-cell origin. Blood. 1996 Dec 1;88(11):4265-74. PMID 8943863
- [Background] Melnyk A, Rodriguez A, Pugh WC, Cabannillas F. Evaluation of the Revised European-American Lymphoma classification confirms the clinical relevance of immunophenotype in 560 cases of aggressive non-Hodgkin's lymphoma. Blood. 1997 Jun 15;89(12):4514-20. PMID 9192775
- [Background] Armitage JO, Weisenburger DD. New approach to classifying non-Hodgkin's lymphomas: clinical features of the major histologic subtypes. Non-Hodgkin's Lymphoma Classification Project. J Clin Oncol. 1998 Aug;16(8):2780-95. doi: 10.1200/JCO.1998.16.8.2780. PMID 9704731
- [Background] Ascani S, Zinzani PL, Gherlinzoni F, Sabattini E, Briskomatis A, de Vivo A, Piccioli M, Fraternali Orcioni G, Pieri F, Goldoni A, Piccaluga PP, Zallocco D, Burnelli R, Leoncini L, Falini B, Tura S, Pileri SA. Peripheral T-cell lymphomas. Clinico-pathologic study of 168 cases diagnosed according to the R.E.A.L. Classification. Ann Oncol. 1997 Jun;8(6):583-92. doi: 10.1023/a:1008200307625. PMID 9261528
- [Background] Lopez-Guillermo A, Cid J, Salar A, Lopez A, Montalban C, Castrillo JM, Gonzalez M, Ribera JM, Brunet S, Garcia-Conde J, Fernandez de Sevilla A, Bosch F, Montserrat E. Peripheral T-cell lymphomas: initial features, natural history, and prognostic factors in a series of 174 patients diagnosed according to the R.E.A.L. Classification. Ann Oncol. 1998 Aug;9(8):849-55. doi: 10.1023/a:1008418727472. PMID 9789607
- [Background] Savage KJ, Chhanabhai M, Gascoyne RD, Connors JM. Characterization of peripheral T-cell lymphomas in a single North American institution by the WHO classification. Ann Oncol. 2004 Oct;15(10):1467-75. doi: 10.1093/annonc/mdh392. PMID 15367405
- [Background] Gallamini A, Stelitano C, Calvi R, Bellei M, Mattei D, Vitolo U, Morabito F, Martelli M, Brusamolino E, Iannitto E, Zaja F, Cortelazzo S, Rigacci L, Devizzi L, Todeschini G, Santini G, Brugiatelli M, Federico M; Intergruppo Italiano Linfomi. Peripheral T-cell lymphoma unspecified (PTCL-U): a new prognostic model from a retrospective multicentric clinical study. Blood. 2004 Apr 1;103(7):2474-9. doi: 10.1182/blood-2003-09-3080. Epub 2003 Nov 26. PMID 14645001
- [Background] Zaja F, Russo D, Silvestri F, Fanin R, Damiani D, Infanti L, Salmaso F, Mariuzzi L, Di Loreto C, Baccarani M. Retrospective analysis of 23 cases with peripheral T-cell lymphoma, unspecified: clinical characteristics and outcome. Haematologica. 1997 Mar-Apr;82(2):171-7. PMID 9175321
- [Background] Tsuchiya T, Ohshima K, Karube K, Yamaguchi T, Suefuji H, Hamasaki M, Kawasaki C, Suzumiya J, Tomonaga M, Kikuchi M. Th1, Th2, and activated T-cell marker and clinical prognosis in peripheral T-cell lymphoma, unspecified: comparison with AILD, ALCL, lymphoblastic lymphoma, and ATLL. Blood. 2004 Jan 1;103(1):236-41. doi: 10.1182/blood-2002-05-1352. Epub 2003 Sep 4. PMID 12958063
- [Result] Federico M, Bellei M, Pesce, E, Zucca E, Pileri S, Montoto S, Weisenburger DD, Ruediger T, KO YH, Liang R, Zinzani PL, Connors JM, Foss FM, Horwitz SM, Polliack A, Vose JM. T-Cell Project: an international, longitudinal, observational study of patients with aggressive peripheral T-cell lymphoma. Revista Brasileira de Hematologia e Hemoterapia 31(suppl 2):21-25,2009.
- [Result] Federico M, Bellei M, Pesce EA, Zucca E, Pielri S, Montoto S, Weisenburger D, Rugiger T, Ko Y, Liang R, Zinzani PL, Connors J, Foss F, Horwitz S, Polliack A, Vose J. T-Cell Project: an international, prospective, observational study of patients with aggressive Peripheral T-cell Lymphoma. Analysis of the first 524 patients. 11 ICML, Lugano (Switzerland), 15-18 June 2011. Abs 241. Ann Oncol 22 (suppl 4), 2011
- [Result] Bellei M, Chiattone CS, Luminari S, Pesce EA, Cabrera ME, de Souza CA, Gabus R, Zoppegno L, Zoppegno L, Milone J, Pavlovsky A, Connors JM, Foss FM, Horwitz SM, Liang R, Montoto S, Pileri SA, Polliack A, Vose JM, Zinzani PL, Zucca E, Federico M. T-cell lymphomas in South america and europe. Rev Bras Hematol Hemoter. 2012;34(1):42-7. doi: 10.5581/1516-8484.20120013. PMID 23049383
- [Result] Federico M, Bellei M, Luminari S, Horwitz SM, Montoto S, Zucca E, Pileri SA, Ko YH, Zinzani PL, Connors JM, Foss FM, Polliack A, Cabrera ME, Kim WS, Spina M, De Souza CA, Bobillo Varela S, Dlouhy I, Advani RH, Vose J and T-Cell Project. CD30+ expression in Peripheral T-cell lymphomas (PTCLs): A subset analysis from the international, prospective T-Cell Project. Journal of Clinical Oncology, 2015 ASCO Annual Meeting (May 29 - June 2, 2015).Vol 33, No 15_suppl (May 20 Supplement), 2015: 8552
- [Result] Federico M, Bellei M, Pesce EA, et al. T-Cell Project: an international, prospective, observational study of patients with aggressive Peripheral NK/T-Cell Lymphoma: Lesson from the first 1308 patients. 13 ICML, Lugano (Switzerland) 17-20 June, 2015. Abstract 070. Hematol Oncol 2015; 33(Suppl1):100-180
- [Result] Bellei M, Marcheselli L, Pesce EA, et al. Clinical Characteristics and Patterns of Care of Patients (pts) with Peripheral T-cell Lymphoma (PTCLs) according to age at time of diagnosis: A T-Cell Project snapshot. 13 ICML, Lugano (Switzerland) 17-20 June, 2015. Abstract 231. Hematol Oncol 2015; 33(Suppl1):181-243
- [Result] Horwitz SM, Bellei M, Marcheselli L, et al. The role of transplant in the treatment of Peripheral T-cell Lymphomas (PTCLs): an analysis from the T-cell Project database. 13 ICML, Lugano (Switzerland) 17-20 June, 2015. Abstract 247. Hematol Oncol 2015; 33(Suppl1):181-243
- [Result] Bellei M, Sabattini E, Pesce EA, Ko YH, Kim WS, Cabrera ME, Martinez V, Dlouhy I, Paes RP, Barrese T, Vassallo J, Tarantino V, Vose J, Weisenburger D, Rudiger T, Federico M, Pileri S. Pitfalls and major issues in the histologic diagnosis of peripheral T-cell lymphomas: results of the central review of 573 cases from the T-Cell Project, an international, cooperative study. Hematol Oncol. 2017 Dec;35(4):630-636. doi: 10.1002/hon.2316. Epub 2016 Jun 3. PMID 27255982
- [Derived] Chiattone C, Civallero M, Fischer T, Miranda E, Manni M, Zing NPC, Pileri SA, Montoto S, Horwitz SM, Cabrera ME, De Souza CA, Nagler A, Luminari S, Ferreri AJM, Carson KR, Re A, Rigacci L, Nassi L, Stepanishyna Y, Federico M, Inghirami G. Characteristics and clinical outcomes of patients with ALK-positive anaplastic large cell lymphoma: Report from the prospective international T-cell lymphoma project. Hematol Oncol. 2022 Dec;40(5):953-961. doi: 10.1002/hon.3074. Epub 2022 Sep 15. PMID 36083035
- [Derived] Advani RH, Skrypets T, Civallero M, Spinner MA, Manni M, Kim WS, Shustov AR, Horwitz SM, Hitz F, Cabrera ME, Dlouhy I, Vassallo J, Pileri SA, Inghirami G, Montoto S, Vitolo U, Radford J, Vose JM, Federico M. Outcomes and prognostic factors in angioimmunoblastic T-cell lymphoma: final report from the international T-cell Project. Blood. 2021 Jul 22;138(3):213-220. doi: 10.1182/blood.2020010387. PMID 34292324
- [Derived] Shustov A, Cabrera ME, Civallero M, Bellei M, Ko YH, Manni M, Skrypets T, Horwitz SM, De Souza CA, Radford JA, Bobillo S, Prates MV, Ferreri AJM, Chiattone C, Spina M, Vose JM, Chiappella A, Laszlo D, Marino D, Stelitano C, Federico M. ALK-negative anaplastic large cell lymphoma: features and outcomes of 235 patients from the International T-Cell Project. Blood Adv. 2021 Feb 9;5(3):640-648. doi: 10.1182/bloodadvances.2020001581. PMID 33560375
- [Derived] Fox CP, Civallero M, Ko YH, Manni M, Skrypets T, Pileri S, Kim SJ, Cabrera ME, Shustov AR, Chiattone CS, Horwitz SM, Dlouhy I, Spina M, Hitz F, Montoto S, Nagler A, Martinez V, De Souza CA, Fernandez-Alvarez R, Ballova V, Gabus R, Inghirami G, Federico M, Kim WS. Survival outcomes of patients with extranodal natural-killer T-cell lymphoma: a prospective cohort study from the international T-cell Project. Lancet Haematol. 2020 Apr;7(4):e284-e294. doi: 10.1016/S2352-3026(19)30283-2. Epub 2020 Feb 24. PMID 32105608
- [Derived] Bellei M, Foss FM, Shustov AR, Horwitz SM, Marcheselli L, Kim WS, Cabrera ME, Dlouhy I, Nagler A, Advani RH, Pesce EA, Ko YH, Martinez V, Montoto S, Chiattone C, Moskowitz A, Spina M, Biasoli I, Manni M, Federico M; International T-cell Project Network. The outcome of peripheral T-cell lymphoma patients failing first-line therapy: a report from the prospective, International T-Cell Project. Haematologica. 2018 Jul;103(7):1191-1197. doi: 10.3324/haematol.2017.186577. Epub 2018 Mar 29. PMID 29599200
- See also: Click here for more information about the T-Cell Project — http://www.tcellproject.org